CLINICAL TRIAL: NCT01968343
Title: Group Treatment for Trichotillomania: Cognitive-Behavioral Therapy Versus Supportive Therapy
Brief Title: Trichotillomania: Group Cognitive-Behavioral Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Hermano Tavares, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CaPPesq 0013/08
Record Dates: First submitted 2013-09-20; First posted 2013-10-24 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2013-10

CONDITIONS: Trichotillomania
MeSH Terms: conditions — Trichotillomania | interventions — Cognitive Behavioral Therapy; Palliative Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Group cognitive-behavioral therapy (Experimental): 22 subjects, all of whom met the criteria for a diagnosis of trichotillomania established in the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition. Subjects receive 22 sessions of group cognitive-behavioral therapy.
  Interventions: Behavioral: Cognitive-behavioral therapy.
- Group supportive therapy (control) (Active Comparator): 22 subjects, all of whom met the criteria for a diagnosis of trichotillomania established in the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition. Subjects receive 22 sessions of group supportive therapy (control).
  Interventions: Other: Supportive therapy.

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy. — Subjects receive 22 sessions of cognitive-behavioral therapy.
  Arms: Group cognitive-behavioral therapy
Other: Supportive therapy. — Subjects receive 22 sessions of supportive therapy.
  Arms: Group supportive therapy (control)

SUMMARY:
Objective: Trichotillomania is a psychiatric condition characterized by chronic pulling and plucking of one's own hair. Cognitive behavioral therapy shows promise as a treatment. However, there have been no randomized, controlled studies of the efficacy of group cognitive-behavioral therapy. Methods: We evaluated 44 subjects, whom met the criteria for a diagnosis of trichotillomania. Subjects were randomized to receive 22 sessions of either group cognitive-behavioral therapy or group supportive therapy (control).

ELIGIBILITY:
Inclusion Criteria:

* Patients having been diagnosed with trichotillomania according to Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV) criteria; being at least 18 years of age; and having had four or more years of schooling.

Exclusion Criteria:

* Patients that having been diagnosed with trichotillomania according to DSM-IV criteria; having less of 18 years of age; and having less of four years of schooling.
* Patients with a history of suicidal ideation,
* Patients with any clinical pathology requiring emergency treatment at admission,
* Patients with mental retardation or any other central nervous system disorder that severely impairs cognitive function,
* those with a psychotic disorder,
* those currently being treated with psychotropic drugs,
* those with any DSM-IV axis II diagnosis,
* those who scored ≤ 2 on the MGH-HPS in an initial screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Massachusetts General Hospital (MGH) Hairpulling Scale (HPS) | 22 weeks
  The MGH-HPS comprises seven self-report items that are scored on a Likert scale (0-4 points).22 Higher MGH-HPS scores correspond to greater severity of trichotillomania symptoms. Reference: Psychotherapy and Psychosomatic Journal 1995;64:141-5

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | 22 weeks
  The BDI consists of 21 items, scored from 0 to 3, higher scores corresponding to greater severity of depression. It is a self-report measure of depression that is widely used in research and in clinical practice. Reference: Archives of General Psychiatry 1961;4:53-63.

OTHER OUTCOMES:
Social Adjustment Scale (SAS) Self-Report (SR) | 22 weeks
  The SAS-SR is a self-report scale consisting of 54 questions addressing seven specific areas in relation to the last two weeks25: work; social life and leisure; family relationships; marital relationship; relationships with children; home life; and financial status, each corresponding to a partial score. Reference: Archives of General Psychiatry 1976;33:111-5.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Psiquiatria da Universidade de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Toledo EL, De Togni Muniz E, Brito AM, de Abreu CN, Tavares H. Group treatment for trichotillomania: cognitive-behavioral therapy versus supportive therapy. J Clin Psychiatry. 2015 Apr;76(4):447-55. doi: 10.4088/JCP.13m08964. PMID 25271779